CLINICAL TRIAL: NCT03758768
Title: The Effects of a Blue Monochromatic Light Intervention on Evening-type Individuals' Sleep and Circadian Rhythms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 271561
Record Dates: First submitted 2018-11-20; First posted 2018-11-29 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Circadian Rhythm Sleep Disorder, Delayed Sleep Phase; Sleep
Keywords: Circadian rhythm; Sleep; evening-type individuals; morningness-eveningness; blue light; monochromatic light; randomized controlled trial
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, single-blinded trial.
Who Masked: Participant, Investigator
Masking Description: A third-party investigator is recruited to be present during the intervention. This third-party investigator has no knowledge of the hypotheses of the study.
  Although the participants can see the type of light they receive, they have no knowledge of the study hypotheses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blue monochromatic light (Experimental): Three consecutive mornings of one hour exposure to monochromatic light (20 lx, irradiance = 49.65 µW/cm2) with peak wavelength of 455 nm (blue light), with equal photon flux as the control condition.
  Interventions: Other: Blue light exposure
- Full spectrum light control condition (Active Comparator): Three consecutive mornings of one hour exposure to full spectrum light (2500 Kelvin, irradiance = 37.72 µW/cm2) with equal photon flux as the blue light.
  We will adjust the light intensity to make sure that the photon energy is the same across the two conditions.
  Interventions: Other: Full spectrum light exposure

INTERVENTIONS:
Other: Blue light exposure — Light administered through ceiling mounted light emitting diode (LED)-based room lighting.
  Arms: Blue monochromatic light
Other: Full spectrum light exposure — Light administered through ceiling mounted light emitting diode (LED)-based room lighting.
  Arms: Full spectrum light control condition

SUMMARY:
The present project is aimed to contribute with new knowledge concerning how light conditions in the physical environment can be manipulated to alter the sleep and circadian rhythms of individuals with an evening-type circadian rhythm. More precisely, the study will explore whether exposure to blue light (compared to a full spectrum light control condition) during the morning hours advance the circadian rhythms of evening-type individuals, towards that which is more similar to the daily rhythm of morning-type individuals. This study is important as it has been found that evening-type adolescents and adults are at higher risk of poor academic performance and demonstrate lower intellectual performance when tested at their nonoptimal early times of day, and given the fact that most schools and workplaces structure their working hours during such early hours of the day. Such an intervention could thus help evening-type individuals better adjust to the different early day requirements that they are exposed to. The project involves a three-day intervention where participants will be exposed to blue monochromatic light, administered through ceiling mounted light emitting diode (LED)-based room lighting, in the early hours of each morning for a duration of 60 min. The participants' sleep, circadian rhythm and waking function will be assessed both objectively and subjectively. The effects of the intervention are transferable to real life educational and work settings and can thus be applied in naturalistic settings. The intervention is based on the new laboratory infrastructure available at the sleep laboratory situated in Christies gate 12.

DETAILED DESCRIPTION:
Background:

Morningness/eveningness is a phenomenon that reflects the tendency to be an "early morning bird" or a "late night owl" and is thus a source of inter-individual variation in timing of sleep and other behaviors. Evening- and morning-type individuals demonstrate differences that derive internally regarding the circadian phase of their endogenous biological clock. A certain group of individuals referred to as morning-type individuals have been consistently found to perform better in the morning, whereas evening-type individuals appear to be more alert and perform better in the evening. Morning-type individuals have earlier bed- and rise times than evening-types, while evening-type individuals have been known to report significantly later bed- and rise-times compared to morning-type individuals. In addition, evening-type adolescents have been known to demonstrate poorer academic and intellectual performances during their nonpreferred, i.e., early hours of the day.

Circadian rhythms are known as biological processes that display endogenous, entrainable oscillations in a period of about 24 hours. These rhythms have been found to be controlled by the circadian pacemaker, which is located in the suprachiasmatic nuclei (SCN) of the hypothalamus. These 24-hour rhythms manifest themselves in an observable manner within numerous physiological measures, such as the sleep-wake cycle, the core body temperature, and the excretion of hormones such as melatonin. The core body temperature falls during the night and reaches its lowest point (nadir) in the early morning, after which it starts to rise again. Melatonin secretion follows a curve which is almost inverse compared to the core body temperature rhythm, and is sensitive to light exposure which inhibits melatonin secretion. Melatonin either in plasma, saliva or urine is regarded as an objective marker of circadian rhythms, of which the dim light melatonin onset (time when melatonin reaches 4 pg/ml in saliva) is the most commonly used parameter.

Sleep is known to be most easily initiated when the core body temperature is falling and as the melatonin level is rising. It is also known to be most easily initiated in a timeframe of six hours before nadir until a couple of hours after nadir of the core body temperature.

Evening-type individuals experience increased sleepiness and poorer performances during the early hours of the morning, as there is a mismatch between their circadian rhythms and their requirement of being awake at such early hours. Sleepiness is known to have severe implications for performance.

However, as mentioned, the SCN outputs are entrainable and light is the strongest time-giver for individuals' circadian pacemakers. Thus, the timing of light exposure has the potential to either phase advance or phase delay one's circadian rhythm. Exposure to light in the hours before nadir, during the evening, will lead to individuals delaying their circadian rhythm. On the other side, exposure to light in the hours after nadir, during the morning hours, has the potential to phase advance individuals' circadian rhythms. Light can shift the circadian phase, but this effect is dependent on the timing of light, duration of light exposure, and the intensity of light where higher intensities have been demonstrated to be associated with greater effects. Another property of light concerns the wavelengths that it emits, where blue light has been shown to produce significantly stronger phase shifting effects than lights of other wavelengths of the visible spectrum. The effects of blue-light on the circadian system has been attributed to a photoresponsive cell population in the retina that contains the photopigment melanopsin, which is highly sensitive to blue light. These cells send signals directly to the SCN, and also form connections to areas associated with wakefulness such as the striatum and the brain stem. The sensitivity to melanopsin has been demonstrated to be highest in a blue light range around 460 nm.

To the best of our knowledge, no study has been conducted to test the effects of a blue monochromatic light intervention administered via standard room lightning on phase advancement of the circadian rhythms of evening-type individuals. Consequently, our aim is to assess whether blue light as compared to standard white light, administered via standard room lightning, can alter the sleep and circadian rhythm of evening-type individuals, causing a phase advance.

Hypothesis:

Three consecutive mornings of one hour exposure to monochromatic light (40 lx, irradiance = 88,79 µW/cm2) with peak wavelength of 455 nm (blue light) will, compared to full spectrum light (2500 Kelvin) with equal photon flux as the blue light: a) lead to a phase advance of the circadian rhythm of evening-type individuals; b) increase waking function assessed with subjective and objective measures in the morning; and c) decrease participants self-reported sleepiness in the morning, d) reduce sleep onset latency and e) advance sleep onset time.

We will adjust the light intensity to make sure that the photon energy is the same across the two conditions.

Methods

Sample and procedure:

Our aim is to recruit a sample of minimum 34 participants from the University of Bergen. Inclusion criteria is scoring below 42 on the Horne-Östberg Morningness-Eveningness Questionnaire, as this categorizes moderate and definitely evening types. Participants will be excluded if a positive case is indicated on the Mood Disorder Questionnaire (MDQ), indicating the presence or history of bipolar disorder. Participants will also be excluded if they have worked night shifts during the past three months. The participants will be exposed to the blue light intervention in a randomized, blinded, controlled study. The participants will be assessed with subjective and objective measures of sleep for 3 days (Tuesday - Thursday) a week before the three-day blue light intervention. They will also be assessed with the same subjective and objective measures during the three-day intervention period. More precisely, sleep will be assessed by actigraphy and sleep diary. One day before the intervention and one day after the intervention, circadian rhythm will be measured by saliva samples for estimation of dim light melatonin onset. Flexibility will also be measured before intervention through the Circadian Type Inventory. Waking function will be assessed on the days the intervention is given with the Karolinska Sleepiness Scale and Psychomotor Vigilance Task.

Instruments/measures:

Circadian Type Inventory: an instrument with two factors. Individuals scoring high on the first dimension (Flexible/Rigid) are more flexible in their ability to stay awake at odd times of day or night. Those who score high on the second factor (Languid/Vigorous) tend to report difficulty in overcoming drowsiness, especially in the morning. CTI will be distributed to participants before the light intervention.

Munich ChronoType Questionnaire: a useful tool for determining chronotype based on sleep behaviors, such as bed- and rise-times, clock time when one becomes fully awake, in addition to some other points (e.g., sleep latency). MCTQ will be distributed to participants before the light intervention.

The Horne-Östberg Morningness-Eveningness Questionnaire (MEQ): a test that has been widely used to assess morningness-eveningness. MEQ will be distributed to participants for screening purposes.

Mood Disorder Questionnaire (MDQ): MDQ is a validated self-report instrument that screens for the presence of a lifetime history of bipolar disorder. It contains 13 yes/no items that cover topics such as mood, self-confidence, energy, sociability, interest in sex, loquaciousness, distractibility, and other behaviors. There are in addition two questions assessing whether the symptoms ever co-occurred and to which degree the symptoms caused functional impairment. A positive case entails endorsement of 7 or more of the 13 symptoms, endorsement of the co-occurrence item and reporting moderate or serious degree of functional impairment. The MDQ will only be administered for screening purposes at baseline.

Actigraphy: Wrist-worn accelerometers and clocks to be worn during the same period as the sleep diary. Data can be converted to objective sleep parameters. This watch will be worn the week before intervention for three days, on the night before Wednesday, Thursday and Friday. It will also be worn in the intervention week on the three intervention days, on the night before Wednesday, Thursday and Friday.

Sleep diary: Daily subjective estimates of bedtime, rise-time, sleep latency, number of awakenings, wake time after sleep onset, final awakening time, rise time, total sleep time, sleep efficiency, sleep quality and daytime functioning.

The questionnaire will be distributed to the participants the week before intervention for three days, on the night before Wednesday, Thursday and Friday. It will also be given in the intervention week on the three intervention days, on the night before Wednesday, Thursday and Friday. Two of the questions are filled before the participants go to bed, and the rest is filled when they wake up in the morning.

Dim light melatonin onset (DLMO): DLMO will be assessed by collecting saliva samples every hour in the evening, starting from 19:00 until one hour after normal bedtime. DLMO samples will be collected one day before the intervention and the day after the intervention period. Saliva collection and analyses will follow procedures previously used by our research group. Blue light blocker glasses will be worn (from one hour prior to the first sample) in order to prevent melatonin suppression during saliva sampling. DLMO will be analyzed with enzyme-linked immunosorbent assay (ELISA) (direct saliva melatonin from Bühlmann Laboratories, Schöonenbuch, Switzerland). The analytical sensitivity of this kit is 0.5 pg/ml and functional sensitivity is 1.6-20.5 pg/ml, with an interassay coefficient of variation of <12.6%. Samples will be analyzed with a Wallac plate reader from Perkin Elmer Inc. (Waltham, MA, USA).

Karolinska Sleepiness Scale (KSS): KSS comprises a single item assessing state sleepiness on a scale from 1 to 9. This instrument will be given in the laboratory on the days of the light intervention. It will be given for a total of six times per participant, twice on each intervention day, the first immediately when the participants come to the laboratory to receive the intervention, and the second after they have received one hour of light, before they leave the laboratory.

Psychomotor Vigilance Task (PVT): a 10-minute reaction-time test that provides a measure of sustained attention will be completed by the participants during light exposure in the laboratory. The participant simply responds to stimuli given on a display by pressing a button as soon as possible. PVT is especially sensitive to sleep loss and fatigue. PVT will be given to participants on the three days of light intervention.

Statistical analysis/power analysis:

A 2 (Time; pre vs post) x 2 (Group; blue vs. full spectrum light) ANOVA will be used for analyzing the results. Power analysis was conducted with G*Power, version 3.17. Setting the effect size to medium (d=0.50), power to .80, alpha to .05, r between repeated measures to .50, shows that 34 participants will be needed in order to detect a significant Time x Group interaction.

ELIGIBILITY:
Inclusion Criteria:

* Scoring below 42 on the Horne-Östberg Morningness-Eveningness Questionnaire, as this categorizes moderate and definitely evening types (Horne & Östberg, 1976).

Exclusion Criteria:

* Participants will be excluded if a positive case is indicated on the Mood Disorder Questionnaire (MDQ), indicating the presence or history of bipolar disorder.
* Participants will also be excluded if they have worked night shifts during the past three months.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2018-10-22 (Actual); Study Completion 2018-10-22 (Actual)

PRIMARY OUTCOMES:
Change scores from baseline to post-intervention in Dim light melatonin onset (DLMO) | Pre-intervention/baseline (Monday in the week of intervention - one day before the first intervention day); Post-intervention (Friday, the week of intervention - one day after last intervention day)
  Melatonin either in plasma, saliva or urine is regarded as an objective marker of circadian rhythms, of which the dim light melatonin onset (time when melatonin reaches 4 pg/ml in saliva) is the most commonly used parameter (Pandi-Perumal et al., 2007).
  The change score of the intervention group will be compared to the change score of the control group. Thus only one parameter will be estimated.
Change scores of Feeling of Morning Wakefulness, measured by Sleep Diary | Tuesday, Wednesday and Thursday (baseline; week before intervention); Tuesday, Wednesday and Thursday (week of light intervention)
  Change scores of the feeling of morning wakefulness across Tuesday to Thursday the week before intervention, substracted from Feeling of Morning Wakefulness across Tuesday to Thursday on the intervention week.
  Since the comparison is made across days/measurement points, only one composite parameter for each condition will be calculated.
Psychomotor Vigilance Task (PVT) | PVT will be given to participants on the three days of light intervention (Tuesday, Wednesday and Thursday). The average score of these three days will be obtained and compared with the control group.
  A 10-minute reaction-time test that provides a measure of sustained attention will be completed by the participants during light exposure in the laboratory. The participant simply responds to stimuli given on a display by pressing a button as soon as possible. PVT is especially sensitive to sleep loss and fatigue (Lamond, Dawson & Roach, 2005).
  Average scores of reaction time across Tuesday, Wednesday and Thursday (the three days of light intervention) will be calculated for the intervention group and compared to the average scores of reaction time across Tuesday, Wednesday and Thursday (the three days of light intervention for the control group.
  Since the comparison is made across days/measurement points, only one composite parameter for each condition will be calculated.
Karolinska Sleepiness Scale (KSS) | Given on the days of intervention (Tuesday, Wednesday, Thursday) twice on each day. First immediately when the participants enter the lab to receive the intervention, and the second after they have received one hour of light, before they leave the lab.
  KSS comprises a single item assessing state sleepiness on a scale from 1 (very rested) to 9 (very sleepy). (Aakerstedt & Gillberg, 1990). The minimum score is 1 (very rested) and the maximum is 9 (very sleepy). Lower values present the feeling of restedness and are thus considered to be a better outcome.
  Average score of KSS will be calculated across the three intervention days (Tuesday, Wednesday, Thursday) for the intervention group, and compared to the average score of KSS across the same three intervention days for the control group. Accordingly, only one outcome measure will be calculated per group. Thus only one parameter will be estimated.

SECONDARY OUTCOMES:
Changes scores in Sleep Length | Change scores of sleep length across Tuesday, Wednesday and Thursday the week before intervention, substracted from sleep length across Tuesday, Wednesday and Thursday on the intervention week.
  Based on sleep diary (subjective measure of sleep length) and actigraphy (objective measure of sleep length).
  The sleep diary consists of no pre-determined scale. It is a diary where the participants fill in a time-point (e.g. the time they went to bed, the time they turned off the lights, how long it took until they fell as asleep, and when they woke up in the morning). The measurement unit is minutes.
  Since the comparison is made across days/measurement points, only one composite parameter for each condition will be calculated.
Change scores in Sleep Onset Time | Change scores of sleep onset time across Tuesday, Wednesday, and Thursday the week before intervention, substracted from sleep onset time across Tuesday, Wednesday, and Thursday on the intervention week.
  Based on sleep diary (subjective measure of sleep onset time) and actigraphy (objective measure of sleep onset time).
  The sleep consists of items that require a time-point as the answer. E.g.: What time did you wake up, to which you can reply 09:00 or any value within a 24-hour day.
  Since the comparison is made across days/measurement points, only one composite parameter for each condition will be calculated.
Changes scores in Wake-up Time | Change scores of wake-up time across Tuesday, Wednesday and Thursday the week before intervention, substracted from wake-up time across Tuesday, Wednesday and Thursday on the intervention week.
  Based on sleep diary (subjective measure of wake-up time) and actigraphy (objective measure of wake-up time).
  The sleep diary consists of items that require a time-point as the answer. E.g.: What time did you wake up, to which you can reply 08:30 or any value within a 24-hour day.
  Since the comparison is made across days/measurement points, only one composite parameter for each condition will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Ståle Pallesen, Principal Investigator — The University of Bergen
Locations (1):
- University of Bergen, Bergen, Hordaland, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Akerstedt T, Gillberg M. Subjective and objective sleepiness in the active individual. Int J Neurosci. 1990 May;52(1-2):29-37. doi: 10.3109/00207459008994241. PMID 2265922
- [Background] Berson DM, Dunn FA, Takao M. Phototransduction by retinal ganglion cells that set the circadian clock. Science. 2002 Feb 8;295(5557):1070-3. doi: 10.1126/science.1067262. PMID 11834835
- [Background] Besoluk S, Onder I, Deveci I. Morningness-eveningness preferences and academic achievement of university students. Chronobiol Int. 2011 Mar;28(2):118-25. doi: 10.3109/07420528.2010.540729. PMID 21231873
- [Background] Bjorvatn B, Pallesen S. A practical approach to circadian rhythm sleep disorders. Sleep Med Rev. 2009 Feb;13(1):47-60. doi: 10.1016/j.smrv.2008.04.009. Epub 2008 Oct 8. PMID 18845459
- [Background] Carney CE, Buysse DJ, Ancoli-Israel S, Edinger JD, Krystal AD, Lichstein KL, Morin CM. The consensus sleep diary: standardizing prospective sleep self-monitoring. Sleep. 2012 Feb 1;35(2):287-302. doi: 10.5665/sleep.1642. PMID 22294820
- [Background] Di Milia, L., Smith, P. A., & Folkard, S. (2005). A validation of the revised circadian type inventory in a working sample. Personality and Individual differences, 39(7), 1293-1305.
- [Background] Do MT, Yau KW. Intrinsically photosensitive retinal ganglion cells. Physiol Rev. 2010 Oct;90(4):1547-81. doi: 10.1152/physrev.00013.2010. PMID 20959623
- [Background] Escribano, C., Díaz-Morales, J. F., Delgado, P., & Collado, M. J. (2012). Morningness/eveningness and school performance among Spanish adolescents: Further evidence. Learning and Individual Differences, 22(3), 409-413.
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Figueiro MG, Bierman A, Rea MS. A train of blue light pulses delivered through closed eyelids suppresses melatonin and phase shifts the human circadian system. Nat Sci Sleep. 2013 Oct 4;5:133-41. doi: 10.2147/NSS.S52203. eCollection 2013. PMID 24124400
- [Background] Goldstein D, Hahn CS, Hasher L, Wiprzycka UJ, Zelazo PD. Time of day, Intellectual Performance, and Behavioral Problems in Morning Versus Evening type Adolescents: Is there a Synchrony Effect? Pers Individ Dif. 2007 Feb;42(3):431-440. doi: 10.1016/j.paid.2006.07.008. PMID 17268574
- [Background] Hirschfeld RM, Williams JB, Spitzer RL, Calabrese JR, Flynn L, Keck PE Jr, Lewis L, McElroy SL, Post RM, Rapport DJ, Russell JM, Sachs GS, Zajecka J. Development and validation of a screening instrument for bipolar spectrum disorder: the Mood Disorder Questionnaire. Am J Psychiatry. 2000 Nov;157(11):1873-5. doi: 10.1176/appi.ajp.157.11.1873. PMID 11058490
- [Background] Horne JA, Ostberg O. A self-assessment questionnaire to determine morningness-eveningness in human circadian rhythms. Int J Chronobiol. 1976;4(2):97-110. PMID 1027738
- [Background] Horne JA, Ostberg O. Individual differences in human circadian rhythms. Biol Psychol. 1977 Sep;5(3):179-90. doi: 10.1016/0301-0511(77)90001-1. PMID 922076
- [Background] Kaida K, Takahashi M, Akerstedt T, Nakata A, Otsuka Y, Haratani T, Fukasawa K. Validation of the Karolinska sleepiness scale against performance and EEG variables. Clin Neurophysiol. 2006 Jul;117(7):1574-81. doi: 10.1016/j.clinph.2006.03.011. Epub 2006 May 6. PMID 16679057
- [Background] Kerkhof GA. Inter-individual differences in the human circadian system: a review. Biol Psychol. 1985 Mar;20(2):83-112. doi: 10.1016/0301-0511(85)90019-5. PMID 3888298
- [Background] Kerkhof GA, Van Dongen HP. Morning-type and evening-type individuals differ in the phase position of their endogenous circadian oscillator. Neurosci Lett. 1996 Nov 8;218(3):153-6. doi: 10.1016/s0304-3940(96)13140-2. PMID 8945751
- [Background] Khalsa SB, Jewett ME, Cajochen C, Czeisler CA. A phase response curve to single bright light pulses in human subjects. J Physiol. 2003 Jun 15;549(Pt 3):945-52. doi: 10.1113/jphysiol.2003.040477. Epub 2003 Apr 25. PMID 12717008
- [Background] Lamond N, Dawson D, Roach GD. Fatigue assessment in the field: validation of a hand-held electronic psychomotor vigilance task. Aviat Space Environ Med. 2005 May;76(5):486-9. PMID 15892548
- [Background] LeGates TA, Fernandez DC, Hattar S. Light as a central modulator of circadian rhythms, sleep and affect. Nat Rev Neurosci. 2014 Jul;15(7):443-54. doi: 10.1038/nrn3743. Epub 2014 Jun 11. PMID 24917305
- [Background] Pandi-Perumal SR, Smits M, Spence W, Srinivasan V, Cardinali DP, Lowe AD, Kayumov L. Dim light melatonin onset (DLMO): a tool for the analysis of circadian phase in human sleep and chronobiological disorders. Prog Neuropsychopharmacol Biol Psychiatry. 2007 Jan 30;31(1):1-11. doi: 10.1016/j.pnpbp.2006.06.020. Epub 2006 Aug 1. PMID 16884842
- [Background] Preckel, F., Lipnevich, A. A., Schneider, S., & Roberts, R. D. (2011). Chronotype, cognitive abilities, and academic achievement: A meta-analytic investigation. Learning and Individual Differences, 21(5), 483-492.
- [Background] Rajaratnam SM, Arendt J. Health in a 24-h society. Lancet. 2001 Sep 22;358(9286):999-1005. doi: 10.1016/S0140-6736(01)06108-6. PMID 11583769
- [Background] Randler, C., & Frech, D. (2006). Correlation between morningness-eveningness and final school leaving exams. Biological Rhythm Research, 37(3), 233-239.
- [Background] Roenneberg T, Wirz-Justice A, Merrow M. Life between clocks: daily temporal patterns of human chronotypes. J Biol Rhythms. 2003 Feb;18(1):80-90. doi: 10.1177/0748730402239679. PMID 12568247
- [Background] Rosenthal L, Day R, Gerhardstein R, Meixner R, Roth T, Guido P, Fortier J. Sleepiness/alertness among healthy evening and morning type individuals. Sleep Med. 2001 May;2(3):243-248. doi: 10.1016/s1389-9457(00)00047-2. PMID 11311688
- [Background] Sasseville A, Paquet N, Sevigny J, Hebert M. Blue blocker glasses impede the capacity of bright light to suppress melatonin production. J Pineal Res. 2006 Aug;41(1):73-8. doi: 10.1111/j.1600-079X.2006.00332.x. PMID 16842544
- [Background] Saxvig IW, Wilhelmsen-Langeland A, Pallesen S, Vedaa O, Nordhus IH, Sorensen E, Bjorvatn B. Objective measures of sleep and dim light melatonin onset in adolescents and young adults with delayed sleep phase disorder compared to healthy controls. J Sleep Res. 2013 Aug;22(4):365-72. doi: 10.1111/jsr.12030. Epub 2013 Jan 30. PMID 23363423
- [Background] Terman, M., & Terman, J. S. (2005). Light therapy. Principles and practice of sleep medicine, 4, 1424-42.
- [Background] Tosini G, Ferguson I, Tsubota K. Effects of blue light on the circadian system and eye physiology. Mol Vis. 2016 Jan 24;22:61-72. eCollection 2016. PMID 26900325
- [Background] Wright HR, Lack LC. Effect of light wavelength on suppression and phase delay of the melatonin rhythm. Chronobiol Int. 2001 Sep;18(5):801-8. doi: 10.1081/cbi-100107515. PMID 11763987